CLINICAL TRIAL: NCT01122251
Title: A Multicenter, Randomized, Parallel Group, Double Blind, Double Dummy Phase II Trial to Evaluate the Efficacy and Safety of the Combinations of Lercanidipine and Valsartan in Comparison to Each Component Administered Alone and to Determine the Optimal Dose Combinations in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Lercanidipine and Valsartan in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Kim, Sung Il / Assistant Manager, Clinical Trial 1 Team
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ZVCL001
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Essential Hypertension
Keywords: hypertension; lercanidipine; valsartan
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — lercanidipine; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lercanidpine + Valsartan (Experimental): L10/V80, L20/V80, L10/V160, L20/V160
  Interventions: Drug: Lercanidipine + Valsartan
- Lercanidipine or Valsartan (Active Comparator): L10, L20, V80, V160
  Interventions: Drug: Lercanidipine or Valsartan
- Placebo (Placebo Comparator): Placebo comparators of Lercanidipine and Valsartan
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lercanidipine + Valsartan — L10/V80, L20/V80, L10/V160, L20/V160
  Arms: Lercanidpine + Valsartan
Drug: Lercanidipine or Valsartan — L10, L20, V80, V160
  Arms: Lercanidipine or Valsartan
Drug: Placebo — Placebo of Lercanidipine and Valsartan
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fixed combination of lercanidipine (10 mg or 20 mg) and valsartan (80 mg or 160 mg), lercanidipine and valsartan alone in reducing blood pressure. The study will investigate the dose response relationship for the combinations and monotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 75
* Essential hypertension at screening (-3 week)

Randomization Criteria:

* Essential hypertension at baseline (90mmHg≤sitDBP≤109mmHg, except sitSBP≥180)

Exclusion Criteria:

* Mean sitDBP≥110mmHg or sitSBP≥180
* Secondary hypertension or suspected secondary hypertension
* Uncontrolled diabetes
* Severe heart disease or severe cerebrovascular disease
* clinically significant hematological test results, renal disease (serum creatinine) or liver disease (ALT or AST)
* History of malignant disease
* Autoimmune disease
* Women with a positive pregnancy test result, breast feeding or intention of pregnancy during the trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
sitDBP | Baseline, Week 8
  Average changes from baseline in sitDBP

SECONDARY OUTCOMES:
sitDBP | Week 4, 8
  Response rates (proportion of patients sitDBP<90mmHg or ≥10-mmHg reduction from baseline)
sitDBP | Week 4
  Average changes from baselin in sitDBP
sitSBP | Week 4, 8
  Average changes from baselini in sitSBP

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - 23 sites in Korea, Seoul, Busan Etc.

REFERENCES:
- See also: High Blood Pressure — http://www.nlm.nih.gov/medlineplus/highbloodpressure.html
- See also: Lercanidipine — http://www.mims.co.uk/Drugs/cardiovascular-system/hypertension/zanidip/
- See also: Valsartan — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0137862534&QV1=VALSARTAN